CLINICAL TRIAL: NCT02182115
Title: Effectiveness of Screening and Decolonization of S. Aureus in Surgery Outpatients
Brief Title: S. Aureus Screening and Decolonization
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1R03HS022912-01 (AHRQ); 1R03HS022912-01 (AHRQ)
Record Dates: First submitted 2014-07-01; First posted 2014-07-08 (Estimated); Results first posted 2017-11-17 (Actual); Last update posted 2019-11-05 (Actual); Status verified 2019-11

CONDITIONS: Wound Infection Due to Staphylococcus Aureus; MRSA Infection of Postoperative Wound
Keywords: Staphylococcus aureus infection; Decolonization; Surgical site infection
MeSH Terms: conditions — Staphylococcal Infections; Surgical Wound Infection | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- standard of care (Active Comparator): Surgeon's routine for preoperative showering.
  Interventions: Drug: standard of care
- antiseptic bundle (Experimental): Patients to use study bundle for 5 days prior to scheduled surgery with the following medications to use at home.
  1. Chlorhexidine gluconate soap applied for bathing daily.
  2. Chlorhexidine gluconate mouthrinse used to rinse mouth twice daily.
  3. Nasal mupirocin to applied inside nostrils twice daily.
  Interventions: Drug: antiseptic bundle

INTERVENTIONS:
Drug: antiseptic bundle — 1. Chlorhexidine gluconate liquid soap for bathing daily.
  2. Chlorhexidine gluconate mouthrinse to use twice daily.
  3. Nasal mupirocin to apply twice daily.
  Other Names: Medications applied at home by patient for 5 days.
  Arms: antiseptic bundle
Drug: standard of care — Surgeon's instructions may include advising patients to use an antiseptic soap prior to surgery.
  Other Names: Follow surgeon's instructions for pre-operative bathing.
  Arms: standard of care

SUMMARY:
Staphylococcus aureus (SA) healthcare-associated infections (HAI) cause significant morbidity and mortality. SA causes 15% of all HAI and 30% of surgical site infections (SSIs). Each year over 40 million Americans undergo operations, 1-10% of whom will acquire SSIs. Such infections double the length of hospitalization and risk of dying, and increase U.S. health care costs by $5-10 billion/year. We need effective interventions to prevent SSIs caused by either methicillin-susceptible (MSSA) or methicillin-resistant (MRSA) strains. Nasal carriers of SA (25-30% of adults) have a 2-14 times greater risk than non-carriers of acquiring an SA SSI. A potential prevention approach is routine pre-operative screening of patients, followed by decolonization of identified SA carriers.

DETAILED DESCRIPTION:
The long term goal of this research is to help reduce the incidence of SSIs caused by SA, both MSSA and MRSA strains. This will help improve the safety and effectiveness of health care for Americans. Achievement of this goal requires that we first address the following critical knowledge gaps: (i) which surgical patients should be screened pre-operatively; (ii) which body site(s) should be screened for optimal SA detection, and (iii) which decolonization approach is optimal for outpatient use. The goal of this study is to conduct the research needed to determine pre-operative SA carriage rates (including by strain type and site of carriage), to evaluate the practicality (adherence, cost) of a SA decolonization protocol that is self-administered by patients at home. We are conducting randomized clinical trial (RCT) of the efficacy of nasal mupirocin ointment, chlorhexidine gluconate (CHG) mouth rinse, and CHG pre-operative bathing, as performed by the patient at home for 5 days pre-operatively. This protocol will be compared with the current standard of care, usually 1-2 showers with an antiseptic soap before the procedure. Briefly, the aims are as follows:

Aim 1: Determine the efficacy of a novel decolonization protocol, compared with standard of care, for eradicating SA carriage pre-operatively in surgery out-patients. We hypothesize that the SA eradication rate will be 2-3 times higher in the intervention arm compared with the standard of care arm.

Aim 2: Obtain data to inform sample size calculations and cost estimates for a future trial to prevent SSIs, determine screening requirements, and assess treatment adherence. We will: determine the proportion of pre-operative patients who are SA carriers and the sites of carriage, by SA type, determine adherence to the study intervention and standard of care, reasons for non-compliance, and gather cost data to provide preliminary evidence of potential cost-effectiveness of the intervention.

Aim 3: Identify risk factors (demographic, medical) for SA carriage. Gather preliminary data on SSIs in study subjects.

ELIGIBILITY:
Inclusion Criteria:

* All patient who are 18 years and older, able to give informed consent and willing to complete the study decolonization protocol.
* Surgery must be scheduled 2 weeks in the future to allow completion of the study protocol prior to the scheduled operation.
* Patients will be admitted from home the day of the surgery or have the surgery done on an outpatient basis.

Exclusion Criteria:

* Currently on antibiotic therapy, allergy to mupirocin or CHG.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2014-07; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan E Kline, MD, MPH, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota Medical Center, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No
Aggregate data will be reported once the study has been completed.

REFERENCES:
- [Derived] Kline SE, Neaton JD, Lynfield R, Ferrieri P, Kulasingam S, Dittes K, Glennen A, Jawahir S, Kaizer A, Menk J, Johnson JR. Randomized controlled trial of a self-administered five-day antiseptic bundle versus usual disinfectant soap showers for preoperative eradication of Staphylococcus aureus colonization. Infect Control Hosp Epidemiol. 2018 Sep;39(9):1049-1057. doi: 10.1017/ice.2018.151. Epub 2018 Jul 24. PMID 30037355

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Standard of Care | Antiseptic Bundle
Started | 53 | 57
Completed | 53 | 57
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Standard of Care: Surgeon's routine for preoperative showering. Surgeon's instructions may include advising patients to use an antiseptic soap prior to surgery.
  Other Name: Follow surgeon's instructions for pre-operative bathing.
- Antiseptic Bundle: Patients to use study bundle for 5 days prior to scheduled surgery with the following medications to use at home.
  Chlorhexidine gluconate soap applied for bathing daily. Chlorhexidine gluconate mouthrinse used to rinse mouth twice daily. Nasal mupirocin to applied inside nostrils twice daily.
- Total: Total of all reporting groups
Arm/Group | Standard of Care | Antiseptic Bundle | Total
Number analyzed (Participants) | 53 | 57 | 110
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 41 | 39 | 80
  >=65 years | 12 | 18 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.5 (13.1) | 58.8 (13.3) | 55.8 (13.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 31 | 53
  Male | 31 | 26 | 57
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 44 | 51 | 95
  Other racial/ethnic groups | 8 | 3 | 11
  Unknown or incomplete racial/ethnic group | 1 | 3 | 4
Staphylococcus aureus carriage [Count of Participants; unit: Participants] | 53 | 57 | 110
STAPHYLOCOCCUS AUREUS TYPE [Count of Participants; unit: Participants]
  Methicillin sensitive Staphylococcus aureus (MSSA) | 48 | 51 | 99
  Methicillin resistant Staphylococcus aureus (MRSA) | 5 | 6 | 11

OUTCOME MEASURES:

1. Primary Outcome: Eradication of Staphylococcus Aureus (SA) Carriage at All 4 Body Sites Tested.
Description: Participants with no SA post-treatment, proportion (%) of participants in each study arm that had no SA detected on the post-treatment cultures from the 4 body sites sampled with swab cultures.
Time Frame: Immediately prior to surgery patients are swabbed again at the 4 body sites to see if SA is present or not.
Measure: Count of Participants; unit: Participants
Groups:
- Antiseptic Bundle: Patients to use study bundle for 5 days prior to scheduled surgery with the following medications to use at home.
  1. Chlorhexidine gluconate soap applied for bathing daily.
  2. Chlorhexidine gluconate mouthrinse used to rinse mouth twice daily.
  3. Nasal mupirocin to applied inside nostrils twice daily.
  antiseptic bundle: 1. Chlorhexidine gluconate liquid soap for bathing daily. 2. Chlorhexidine gluconate mouthrinse to use twice daily. 3. Nasal mupirocin to apply twice daily.
Arm/Group | Standard of Care | Antiseptic Bundle
Number analyzed (Participants) | 53 | 57
Participants | 13 | 41

ADVERSE EVENTS:
Time Frame: 2 years
Groups:
- Standard of Care: Used surgeon recommended soap for two pre-op showers, one the night before and one the morning of surgery.
- Antiseptic Bundle: Used three drug antiseptic bundle for 5 days.
Arm/Group | Standard of Care | Antiseptic Bundle
All-Cause Mortality (participants affected / at risk) | 0/53 | 0/57
Serious Adverse Events (participants affected / at risk) | 4/53 | 10/57
Other Adverse Events (participants affected / at risk) | 0/53 | 0/57
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard of Care (N=53) | Antiseptic Bundle (N=57)
non-healing wound (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
pulmonary embolus (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
radial nerve palsy (Nervous system disorders) | 1 (1) | 0 (0)
DVT (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
UTI (Renal and urinary disorders) | 1 (1) | 1 (1)
bacteremia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
lung collapse (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
subdural hematoma (Nervous system disorders) | 0 (0) | 1 (1)
post-op pseudomeningocele (Nervous system disorders) | 0 (0) | 1 (1)
thoracic spine fracture post-op (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
uncontrolled post-operative pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Chyle leak (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
swallowing difficulties (Gastrointestinal disorders) | 0 (0) | 1 (1)
cervical seroma (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
gross hematuria (Renal and urinary disorders) | 0 (0) | 2 (2)
Clostridium difficile diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Limitations include the small number of participants with methicillin resistant SA (MRSA) and with SA carriage at non-nares sites. We were unable to assess the decolonization bundle's efficacy for MRSA and for sites other than nares and perianal.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No